CLINICAL TRIAL: NCT06147544
Title: A Single Center, Randomized, Double Blind, Placebo Controlled, Multiple Dose Escalating Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PB-718 Injection in Chinese Obese Subjects.
Brief Title: A Study to Evaluate the Safety, Tolerability, and Pharmacokinetics of PB-718 Injection in Chinese Obese Subjects.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: PegBio Co., Ltd. (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: PB718101
Record Dates: First submitted 2023-08-09; First posted 2023-11-27 (Actual); Last update posted 2024-04-19 (Actual); Status verified 2024-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PB-718 (Experimental): Low dose level of PB-718 administered on the first day of week 1-12(for cohort 1 and 2) or week 1-18(for cohort 3) according to the dose-escalation design
  Medium dose level of PB-718 administered on the first day of week 1-12(for cohort 1 and 2) or week 1-18(for cohort 3) according to the dose-escalation design
  High dose level of PB-718 administered on the first day of week 1-12(for cohort 1 and 2) or week 1-18(for cohort 3) according to the dose-escalation design
  Interventions: Drug: PB-718
- Placebo (Placebo Comparator): Matched placebo administered on the first day of week 1-12(for cohort 1 and 2) or week 1-18(for cohort 3) according to the dose-escalation design
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: PB-718 — Administered subcutaneously once a week
  Arms: PB-718
Drug: Placebo — Administered subcutaneously once a week
  Arms: Placebo

SUMMARY:
The trial is conducted in a single center, randomized, double blind, placebo controlled, dose increasing design. To evaluate the safety, tolerability, pharmacokinetics(PK) characteristics, efficacy and immunogenicity of PB-718 injection in Chinese obese subjects.

DETAILED DESCRIPTION:
The trial is conducted in a single center, randomized, double blind, placebo controlled, dose increasing design. To evaluate the safety, tolerability, PK characteristics, efficacy and immunogenicity of PB-718 injection in Chinese obese subjects. The study consists of three dose groups, each of which is planned to include 12 subjects (9 receiving the study drug and 3 receiving placebo), for a total of 36 patients. Subjects will receive 12 weeks（for cohort 1 and 2） or 18 weeks(for cohort 3) of treatment after screening and complete 8 weeks of safety follow-up.

ELIGIBILITY:
Inclusion Criteria:

1. Chinese male or female subjects aged 18-60 years (both inclusive).
2. Body weight ≥70 kg(male) or 60 kg(female), and body mass index (BMI) ≥28.0 kg/m2 at screening.
3. Weight change <5% in the past 3 months before screening.

Exclusion Criteria:

1. FPG ≥7.0mmol/L or glycosylated hemoglobin (HbA1c) ≥6.5% or diagnosed diabetes
2. FPG <3.9 mmol/L at screening and/or a history of hypoglycemia.
3. History of Cushing's syndrome, polycystic ovaries, or other hereditary endocrine disorders, or obesity caused by secondary factors such as cortisol hormones.
4. Abnormal Thyroid-Stimulating Hormone(TSH), free triiodothyronine(FT3), Free thyroxine(FT4) or diagnosed thyroid dysfunction
5. History of multiple endocrine neoplasia syndrome type 2 (MEN-2) or medullary thyroid carcinoma (MTC).
6. Diagnosed cardiovascular and cerebrovascular diseases with obvious clinical significance within 6 months before screening
7. Systolic blood pressure > 160 mmHg and/or diastolic blood pressure > 100 mmHg at screening or randomization.
8. PR intervals > 210 msec and/or QRS wave group time limit > 120 msec and/or Corrected QT interval using Fridericia's formula（QTcF）> 450 msec at screening or randomization.
9. Serum amylase or lipase > 3× upper limit of normal (ULN) at screening or before randomization, or previously diagnosed acute/chronic pancreatitis.
10. Low density lipoprotein cholesterol(LDL-C) ≥4.40 mmol/L or triglyceride (TG) ≥5.65 mmol/L.
11. Use of any approved or unapproved drugs or products that have an effect on body weight within 3 months prior to screening
12. History of bariatric surgery for weight loss 1 year before screening.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2023-07-06 (Actual); Primary Completion 2024-04-16 (Actual); Study Completion 2024-04-16 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | From the first dosing (Day 1 ) of study drug until completion of the post treatment follow-up visit (20 weeks for cohort 1 and cohort 2 or 26 weeks for cohort 3)

SECONDARY OUTCOMES:
Pharmacokinetic profile | From the first dose (Day 1 ) of study drug until week 12 (for cohort 1 and cohort 2) or week 18(for cohort 3)
  Cmax
Pharmacokinetic profile | From the first dose (Day 1 ) of study drug until week 12(for cohort 1 and cohort 2) or week 18(for cohort 3)
  Tmax
Pharmacokinetic profile | From the first dose (Day 1 ) of study drug until week 12(for cohort 1 and cohort 2) or week 18(for cohort 3)
  Area under the concentration-time curve over dosing interval(AUC0-tau）
Pharmacokinetic profile | From the first dose (Day 1 ) of study drug until week 12(for cohort 1 and cohort2) or week 18(for cohort 3)
  Area under the concentration-time curve from time zero to the time of the last quantifiable concentration（AUC0-last）
Pharmacokinetic profile | From the first dose (Day 1 ) of study drug until week 12(for cohort 1 and cohort 2) or week 18(for cohort3)
  t1/2
Proportion of participants with ≥5% weight loss | week 12 (for cohort 1 and cohort2) or week 18(for cohort 3)
Change in body weight from baseline | Week12(for cohort 1 and cohort 2) or week 18(for cohort 3)
Change in Fasting Plasma Glucose(FPG) from baseline | week 12(for cohort 1 and cohort 2) or week 18(for cohort 3)

CONTACTS AND LOCATIONS:
Overall Officials: Dongyang liu, PhD, Principal Investigator — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No